CLINICAL TRIAL: NCT05556720
Title: Bringing Optimised COVID-19 Vaccine Schedules To ImmunoCompromised Populations (BOOST-IC): an Adaptive Randomised Controlled Clinical Trial
Acronym: BOOST-IC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: The University of Sydney, Sydney, Australia (Unknown); University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 122.22
Record Dates: First submitted 2022-08-23; First posted 2022-09-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: HIV; Organ Transplantation; Lymphoma, Non-Hodgkin; Chronic Lymphocytic Leukemia; Multiple Myeloma; COVID-19 Vaccines
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma | interventions — BNT162b5; Spikevax bivalent zero omicron; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Intervention Model Description: Study participants who have received three to eight doses of Australian TGA approved COVID-19 vaccine will be randomised into one of up to three groups. They will be administered either one or two homologous doses of COVID-19 vaccines, e.g. Moderna mRNA vaccine OR Pfizer mRNA vaccine, using a central computer-generated random allocation algorithm, with random block sizes of 3 or 6.
  Randomisation will be stratified by:
  - Study subgroup (HIV, solid organ transplant, haematological malignancy)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both study participants and investigators will be blinded to treatment allocation. Individual assignments will be delivered securely and confidentially to the identified site personnel administering the vaccines via a web-based portal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- People living with Human Immunodeficiency Virus (HIV) (Experimental): Eligible participants living with HIV will be randomised 1:1:1 to receive a one or two doses of either current TGA approved COVID-19 vaccines
  1. Moderna COVID-19 vaccine, SPIKEVAX XBB1.5 Adult dose of Spikevax XBB.1.5 contains 50 micrograms of messenger ribonucleic acid (mRNA) (Andusomeran) that encodes the spike protein of the XBB.1.5 strain of the virus.
  2. PfizerCOVID-19 vaccine, COMIRNATYOMICRONXBB.1.5 Adult dose of Comirnaty Omicron XBB.1.5 contains 30 micrograms of a single-stranded, 5'-capped messenger RNA (mRNA) (Raxtozinameran) which encodes the spike protein of the XBB.1.5 strain of the virus.
  Interventions: Biological: Pfizer Bivalent COVID-19 Vaccine; Biological: Moderna Bivalent mRNA vaccine
- Solid Organ Transplant recipients (Experimental): Eligible participants who have previously received at least one solid organ transplant, including kidney, pancreas, liver, heart, lung, or any combination of these organs at least 6 weeks prior and without episodes of severe rejection requiring T- or B-cell depleting agents in the prior 3 months, will be randomised 1:1:1 to receive a one or two doses of bivalent COVID-19 vaccine:
  1. Moderna bivalent COVID-19 vaccine, SPIKEVAX BIVALENT ORIGINAL/OMICRON BA.4-5 (elasomeran/davesomeran); 25 micrograms of imelasomeran that targets the Omicron variant BA.4-5, and 25 micrograms of elasomeran that targets the ancestral strain of SARSCoV-2.
  2. Pfizer bivalent COVID-19 vaccine, COMIRNATY ORIGINAL/OMICRON BA.4-5 (tozinameran/famtozinameran); 15 µg of tozinameran and 15 µg of famtozinameran.
  3. TBC
  Interventions: Biological: Pfizer Bivalent COVID-19 Vaccine; Biological: Moderna Bivalent mRNA vaccine
- People with Haematological Neoplasms (CLL, NHL, MM) (Experimental): Undergoing chemotherapy, immunotherapy and/or targeted therapy, or completed in the last 2 years for chronic lymphocytic leukemia, multiple myeloma or non-Hodgkin lymphoma will be randomised 1:1:1 to receive a one or two doses of bivalent COVID-19 vaccine:
  1. Moderna bivalent COVID-19 vaccine, SPIKEVAX BIVALENT ORIGINAL/OMICRON BA.4-5 (elasomeran/davesomeran); 25 micrograms of imelasomeran that targets the Omicron variant BA.4-5, and 25 micrograms of elasomeran that targets the ancestral strain of SARSCoV-2.
  2. Pfizer bivalent COVID-19 vaccine, COMIRNATY ORIGINAL/OMICRON BA.4-5 (tozinameran/famtozinameran); 15 µg of tozinameran and 15 µg of famtozinameran.
  3. TBC
  Interventions: Biological: Pfizer Bivalent COVID-19 Vaccine; Biological: Moderna Bivalent mRNA vaccine

INTERVENTIONS:
Biological: Pfizer Bivalent COVID-19 Vaccine — One or Two doses three months apart, per manufacturer's recommendations.
  Other Names: Pfizer-BioNTech bivalent mRNA vaccine; COMIRNATY Original/Omicron BA.1
Biological: Moderna Bivalent mRNA vaccine — One or Two doses three months apart, per manufacturer's recommendations.
  Other Names: Moderna Bivalent Original/Omicron; Elasomeran/imelasomeran; Spikevax

SUMMARY:
Despite the greater risk of adverse COVID-19 outcomes, antibody and cell-mediated immune responses to COVID-19 vaccines vary amongst immunocompromised (IC) people and are poorly defined. IC hosts were largely excluded from the COVID-19 vaccine registration trials, though many countries recommend additional and booster doses of vaccination in this group.

BOOST-IC is an adaptive randomised clinical trial (RCT) to assess the immunogenicity and safety of additional COVID-19 vaccine doses in immunocompromised (IC) people, including people with HIV, solid organ transplants (SOT) recipients or those with haematological malignancies. Briefly, the study aims to generate high-quality evidence on the immunogenicity and safety of alternative COVID-19 booster strategies against SARS-CoV-2 for IC people in Australia.

DETAILED DESCRIPTION:
Despite the greater risk of adverse COVID-19 outcomes, antibody and cell-mediated immune responses to COVID-19 vaccines vary amongst immunocompromised (IC) people and are poorly defined. IC hosts were largely excluded from the COVID-19 vaccine registration trials, though many countries recommend additional and booster doses of vaccination in this group. However, data are heterogeneous, in part due the variable nature of immunodeficiencies in IC groups and non-standardised outcome measures used in studies.

BOOST-IC is an adaptive randomised clinical trial (RCT) to assess the immunogenicity and safety of additional bivalent COVID-19 vaccine doses in immunocompromised (IC) people, including people with HIV, solid organ transplants (SOT) recipients or those with haematological malignancies. Briefly, the study aims to generate high-quality evidence on the immunogenicity and safety of alternative COVID-19 booster strategies against SARS-CoV-2 for IC people in Australia.

To do this, participants who have previously completed 3- to 8-doses of Australian TGA approved COVID-19 vaccines (Moderna and Pfizer vaccines) will be randomised 1:1 to receive either one or two doses of the current TGA approved COVID-19 vaccine. .An additional arm can be added if an additional suitable vaccine becomes available. Namely, patients will be randomised to receive either one or two doses of Moderna or Pfizer COVID-19 vaccine. As additional COVID-19 vaccines become available in Australia, these will be included in the trial, as additional arms. The trial can incorporate up to three arms at one time.

Patients will be followed up for 455 days post randomisation. Specific study questions pertain to:

* examining how additional doses of COVID-19 vaccine/s affect correlates of protective immunity
* examining the safety of additional doses of COVID-19 vaccine/s
* characterising the humoral and cellular immune responses to COVID-19 vaccination receiving 1 or 2 booster doses of COVID-19 vaccine/s

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent and undertake study procedures
* Age ≥16 years old
* Have completed at least 3 months prior, 3- to 8-doses of an Australian TGA approved SARS-CoV-2 vaccine (including mRNA [Pfizer or Moderna], ChAdOx1 [Oxford/Astra Zeneca] or protein [Novavax])
* Fit the criteria to be included in one of the following 3 populations: Infected with HIV; Current recipient of a solid organ transplant including: kidney, pancreas, liver, malignancy episodes of severe rejection requiring T- or B-cell depleting agents in the prior 3 months; Undergoing chemotherapy, immunotherapy and/or targeted therapy, or completed in the last 2 years for: chronic lymphocytic leukemia, multiple myeloma or non-Hodgkin lymphoma.

Exclusion Criteria:

* Are contraindicated to receive a COVID-19 booster vaccination, e.g. history of anaphylaxis to a vaccine component or myocarditis attributed to previous receipt of an mRNA vaccine.
* Has had less than 3 or more than 8 doses of COVID-19 vaccine
* Is on another clinical trial investigating alternate COVID-19 vaccination schedules or investigational drugs to prevent or treat COVID-19
* Life expectancy < 12 months, or enrolment deemed not in the best interest of the patient
* Unable to provide informed consent
* Receipt of SARS-CoV-2 specific monoclonal antibodies in the 3 months prior to receiving the first dose of study vaccine
* Acute respiratory tract infection and/or temperature > 38 degrees centigrade on day of receiving first dose of study vaccine
* History of autologous stem cell transplant in the prior 6 months or history of ever having an allogeneic stem cell transplant or CAR T-cell therapy
* Have not received another licensed vaccine in the 7 days before or 7 days after the day of receiving the COVID-19 study vaccine (NOTE: Participants can receive another licensed vaccine on the same day as the COVID-19 vaccine)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The geometric mean concentration (GMC) of anti-spike SARS-CoV-2 IgG antibody against SARS-CoV-2 | 28 days after completion of trial vaccine/s
  geometric mean concentration (GMC) of anti-spike SARS-CoV-2 IgG (AU/ml)

SECONDARY OUTCOMES:
anti-Spike IgG antibody geometric mean concentration | Up to 12 months post completion of trial vaccine/s
  The geometric mean concentration (GMC) (AU/ml) of anti-spike SARS-CoV-2 IgG antibody against SARS-CoV-2 6- and 12-months after completion of trial vaccine/s
Seroconversion | 1-, 6- and 12-months after completion of trial vaccine/s
  The proportion of participants seronegative to SARS-CoV-2 IgG becoming seropositive 1-, 6- and 12-months after completion of trial vaccine/s
Neutralisation responses | Up to 12 months post completion of trial vaccine/s
  Proportion of participants with SARS-CoV-2 neutralising antibody response in each group after 1-, 6- and 12-months post completion of trial vaccine/s, with response defined as either 4-fold rise in the neutralising antibody titre for those with detectable neutralising antibodies at baseline, OR Detectable neutralisation in those with no detectable neutralising antibodies at baseline
T cell polyfunctionality | Up to 12 months post completion of trial vaccine/s
  Subset analysis and polyfunctionality (number, and concentration of effector cytokines) of SARS-CoV-2 specific T-cell responses at 1-, 6- and 12-months post completion of trial vaccine/s in a subset of participants.
T lymphocyte responses | Up to 12 months post completion of trial vaccine/s
  Magnitude of SARS-CoV-2 specific T-cell responses at 1-, 6- and 12-months post completion of trial vaccine/s in a subset of participants
Early local and systemic reactions | Up to 7 days post completion of trial vaccine/s
  Local and systemic reactions assessed by questionnaire on Day 1,2,3,4,5,6 and 7 after randomisation.
  Solicited and unsolicited adverse events following immunisation (AEFI) up to Day 28.
  Hospitalisation resulting from adverse events following immunisation (AEFI) up to Day 28.
Adverse Events Following Immunisation | Up to 28 days post completion of trial vaccine/s
  Proportion with solicited and unsolicited adverse events following immunisation (AEFI) up to Day 28.
Hospitalisation due to Immunisation | Up to 28 days post completion of trial vaccine/s
  Proportion of participants with hospitalisation resulting from adverse events following immunisation (AEFI) up to Day 28.
Clinical outcomes - COVID-19 infection | Up to 12 months post completion of trial vaccine/s
  Proportion of patients with PCR-confirmed OR rapid antigen test (RAT) positive SARS-CoV-2 infection in participants up to 12-months post completion of trial vaccine/s
Clinical outcomes - Healthcare Attendance Due to COVID-19 infection | Up to 12 months post completion of trial vaccine/s
  Proportion of participants with PCR-confirmed OR rapid antigen test (RAT) positive SARS-CoV-2 infection requiring attendance at a medical facility for assessment and/or hospital admission up to 12-months post completion of trial vaccine/s
Clinical outcomes - All Cause and SARS-CoV-2 Related Mortality | Up to 12 months post completion of trial vaccine/s
  Proportion of participants experiencing mortality due to i) any cause and ii) SARS-CoV-2 infection up to 12-months post completion of trial vaccine/s
Clinical outcomes - Severity | Up to 12 months post completion of trial vaccine/s
  Proportion of participants needing oxygen therapy and/or ventilatory support due to SARS-CoV-2 infection up to 12-months post completion of trial vaccine/s Need for ICU care due to SARS-CoV-2 infection up to 12-months post completion of trial vaccine/s
Clinical outcomes - Severe COVID-19 | Up to 12 months post completion of trial vaccine/s
  Proportion of Participants with need for ICU care due to SARS-CoV-2 infection up to 12-months post completion of trial vaccine/s
Clinical outcomes - Quality of Life | Up to 12 months post completion of trial vaccine/s
  Quality of life estimates (using EQ-5D-5L survey) at 1-, 6- and 12-months post completion of trial vaccine/s
Clinical outcomes - Healthcare utilisation | Up to 12 months post completion of trial vaccine/s
  Proportion of participants with healthcare utilisation including outpatient pharmaceutical and medical service use and inpatient hospital admissions related to COVID-19 or study vaccines up to 12-months post completion of trial vaccine/s
Clinical outcomes - All cause healthcare utilisation | Up to 12 months post completion of trial vaccine/s
  Proportion of participants with healthcare utilisation including outpatient pharmaceutical and medical service use and inpatient hospital admissions

CONTACTS AND LOCATIONS:
Overall Officials: James H McMahon, MBBS PhD, Principal Investigator — Alfred Hospital, Melbourne, Australia
Locations (13):
- Australia (13):
  - St Vincents Hospital, Darlinghurst, New South Wales
  - Prince Of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St Vincents Hospital, Fitzroy, Victoria
  - University Geelong Hospital, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Alfred Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dymock M, McMahon JH, Griffin D, Hagenauer M, Snelling TL, Marsh JA; On behalf of the BOOST-IC Investigator Team. Bringing optimised COVID-19 vaccine schedules to immunocompromised populations: statistical elements and design. Trials. 2025 Jul 25;26(1):256. doi: 10.1186/s13063-025-08965-w. PMID 40713834
- [Derived] Zorger AM, Hirsch C, Baumann M, Feldmann M, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with haematological malignancies. Cochrane Database Syst Rev. 2025 May 21;5(5):CD015530. doi: 10.1002/14651858.CD015530.pub2. PMID 40396505
- [Derived] Griffin DWJ, Dymock M, Wong G, Morrissey CO, Lewin SR, Cheng AC, Howard K, Marsh JA, Subbarao K, Hagenauer M, Roney J, Cunningham A, Snelling T, McMahon JH. Bringing optimised COVID-19 vaccine schedules to immunocompromised populations (BOOST-IC): study protocol for an adaptive randomised controlled clinical trial. Trials. 2024 Jul 17;25(1):485. doi: 10.1186/s13063-024-08315-2. PMID 39020446